CLINICAL TRIAL: NCT07057778
Title: Iguratimod Plus Low-dose Rituximab vs Low-dose Rituximab in Corticosteroid-resistant or Relapsed ITP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); Navy General Hospital, Beijing (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pku-IGU-ITP-03
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: Iguratimod
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — iguratimod; Rituximab

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned at a 1:1 ratio to receive Iguratimod plus low-dose rituximab or high-dose rituximab alone. Each group requires 60 patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iguratimod plus low-dose rituximab (Experimental): Low-dose rituximab was used in combination with Iguratimod
  Interventions: Drug: Iguratimod; Drug: low-dose rituximab
- Low-dose rituximab (Active Comparator): Low-dose rituximab alone
  Interventions: Drug: low-dose rituximab

INTERVENTIONS:
Drug: Iguratimod — oral iguratimod at 25mg twice daily for 26 weeks
  Arms: Iguratimod plus low-dose rituximab
Drug: low-dose rituximab — rituximab 100mg once weekly for 6 weeks

SUMMARY:
Randomized, open-label, multicentre study to assess the efficacy and safety of the combination of low-dose rituximab and Iguratimod in patients with steroid-resistant/relapsed ITP.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a severe bleeding disorder. Approximately 2/3 of patients achieve remission from first-line therapies. However, the underlying mechanism of steroid-resistant or relapsed ITP is not well understood; thus, treatment remains a great challenge. Rituximab has been shown to partly improve the complete remission rate of ITP. The small molecule compound iguratimod is widely used as a novel antirheumatic drug to treat several autoimmune diseases. According to studies involving ITP mice, iguratimod may represent a new approach for the prevention and treatment of anti-platelet antibody-mediated ITP by modulating T-cell differentiation.

A multicentre prospective study was performed in non-splenectomized ITP patients who were either resistant to a standard dose of corticosteroids or had relapsed. Patients were randomized to the low-dose rituximab+iguratimod and the low-dose rituximab monotherapy groups. Platelet count, bleeding and other symptoms were evaluated before and after treatment.Adverse events are also recorded throughout the study, in order to assess the efficacy and safety of the combination of low-dose rituximab and iguratimod in patients with steroid-resistant/relapsed ITP.

ELIGIBILITY:
Inclusion Criteria:

* ITP confirmed by excluding other supervened causes of thrombocytopenia;
* Platelet count of less than 30×10^9/L at enrollment;
* Patients who did not achieve a sustained response to treatment with full dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;

Exclusion Criteria:

* Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus);
* Congestive heart failure;
* Severe arrhythmia;
* Nursing or pregnant women;
* Aspartate aminotransferase and alanine transaminase levels ≥ 3×the upper limit of the normal threshold criteria;
* Creatinine or serum bilirubin levels each 1•5 times or more than the normal range;
* Active or previous malignancy;
* Patients with other diseases were undergoing treatment with immunosuppressants;
* Patients with ITP had received rituximab;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
overall response | From the start of study treatment (Day 1) up to the end of Year 1
  The number of participants (responders) with platelet count >=30x10^9/L and at least a 2-fold increase in the baseline count (PR) or a platelet count >=100x10^9/L (CR) and the absence of bleeding, without rescue medication at 1-year follow-up.

SECONDARY OUTCOMES:
sustained response | From the start of study treatment (Day 1) up to the end of Year 1
  The number of participants that can maintain the platelet count > 30 x 109/L, an absence of bleeding events, and without requirement for any other ITP-specific treatment for 6 consecutive months after achievement of response.
complete response | From the start of study treatment (Day 1) up to the end of Year 1
  The number of participants (responders) with platelet count>=100x10^9/L (CR) and the absence of bleeding, without rescue medication at 1-year follow-up.
time to response | From the start of study treatment (Day 1) up to the end of Year 1
  Time to response was defined as the time from starting treatment to the time to achieve the response.
duration of response | From the start of study treatment (Day 1) up to the end of Year 1
  Duration of response was measured from the achievement of response to the loss of response.
incidence of adverse events | All patients were assessed for adverse events every week during the first 4 weeks of treatment, and at 2-weeks interval for the following 5 months, and monthly thereafter. Adverse events were scaled according to CTCAE 5.0
  From the start of study treatment (Day 1) up to the end of Year 1
Bleeding events | From the start of study treatment (Day 1) up to the end of Year 1
  Clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale.
Health-related quality of life (HRQoL) | From the start of study treatment (Day 1) up to the end of Year 1
  ITP-PAQ is used to assess the Health Related Quality of Life (HRQoL) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Beijing, China

IPD SHARING:
Plan to Share IPD: No